CLINICAL TRIAL: NCT04745962
Title: Clinical Evaluation of the Thin TCP-EBUS Bronchoscopy System
Brief Title: Thin EBUS Pilot Study
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Collaborators: Olympus Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 00083498
Record Dates: First submitted 2021-02-04; First posted 2021-02-09 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Lung; Node

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Procedural group
  Interventions: Device: Slimscope

INTERVENTIONS:
Device: Slimscope — Slimscope thin EBUS endoscope is inserted and used to visualize lung nodules.

SUMMARY:
This is a single-center pilot study at the Medical University of South Carolina (MUSC) to evaluate the safety and efficacy of the TCP-EBUS scope (Thin EBUS). This study will consist of a standard of care bronchoscopy and will be followed for approximately 3 months. While the device is not FDA approved, it is the same technology but a thinner version of the SCP-EBUS bronchoscope.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent.
2. >21 years of age or older.
3. Target lesion(s) within the middle third of the lung, which will be determined radiographically prior to scheduling the procedure by the bronchoscopist or radiologist, or by being located at least 2 airway generations from the main carina as seen radiographically.
4. Target lesion(s) location documented on CT scan report.
5. Indicated for bronchosocpy.
6. Bronchoscopic procedure scheduled within 30 days of the CT scan report.

Exclusion Criteria:

1. Not suitable for flexible bronchoscopy as determined by the treating physician prior to the procedure.
2. Currently on anticoagulation medications with INR >1.5.
3. Currently using DOAC and does not suspend use at least 7 days prior to the index procedure
4. Currently using Plavix and does not suspend use for at least 7 days prior to the index procedure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of patients who are scheduled for standard of care assessment of central pulmonary nodules.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2024-09-28 (Actual); Study Completion 2024-09-28 (Actual)

PRIMARY OUTCOMES:
Ability to visualize lung nodule | Throughout the procedure (approximately 1 hour)
  Study team will determine whether or not the lung nodule was able to be visualized by the scope.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas J Pastis, MD, Principal Investigator — The Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No